CLINICAL TRIAL: NCT02253914
Title: An Investigator Blinded, Randomized, Placebo-controlled Multiple Dose Escalation Study of the Safety, Tolerability and Pharmacokinetics of BILR 355 BS Plus Low Dose Ritonavir in HIV-uninfected Male Volunteers
Brief Title: Dose Escalation Study of the Safety, Tolerability and Pharmacokinetics of BILR 355 BS Plus Low Dose Ritonavir in HIV-uninfected Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1188.2
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Solutions; Tablets; Ritonavir

ARMS (3):
- BILR 355 BS, solution (Experimental): escalating doses
  Interventions: Drug: BILR 355 BS, solution; Drug: Ritonavir
- BILR 355 BS, tablet (Experimental): escalating doses
  Interventions: Drug: BILR 355 BS, tablet; Drug: Ritonavir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BILR 355 BS, solution
  Arms: BILR 355 BS, solution
Drug: BILR 355 BS, tablet
  Arms: BILR 355 BS, tablet
Drug: Ritonavir
  Arms: BILR 355 BS, solution; BILR 355 BS, tablet
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to determine the safety, tolerability and pharmacokinetics of BILR 355 BS plus low dose ritonavir in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Males who meet the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
   * No finding deviating from normal (except as noted below) and of clinical relevance
   * No evidence of a clinically relevant concomitant disease
2. Age ≥18 years and <60
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Current and medically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
7. Intake of drugs with a long half-life (>24 hours) within one month prior to administration of study drug or during the trial
8. Use of drugs within 10 days prior to administration or during the trial, which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation
9. Participation in another trial with an investigational drug within one month prior to administration or during the trial
10. Smoker
11. Inability to refrain from smoking on trial days
12. Alcohol abuse (more than 60 g/day)
13. Drug abuse
14. Recent blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
15. Excessive physical activities (within 1 week prior to administration or during the trial)
16. Any laboratory value outside the normal reference range that is of clinical relevance
17. Inability to comply with dietary regimen of study centre
18. Infected with hepatitis B or hepatitis C viruses (defined as either being hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody positive)
19. HIV-1 infected as defined by a positive HIV ELISA test

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2004-02; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
AUCτ (area under the concentration time curve of BILR 355 in plasma over one dosing interval at steady state) | up to day 11
Cmax (maximum concentration of BILR 355 in plasma) | up to day 11
Time for BILR 355 BS to achieve steady state | up to day 11
Cmin,ss (trough concentration of BILR 355 BS in plasma at steady state) | up to day 11
Incidence of dose limiting toxicity | up to day 21

SECONDARY OUTCOMES:
tmax (time from dosing to the maximum concentration of BILR 355 in plasma) | up to day 11
AUCτ (area under the concentration time curve of metabolite 402 in plasma over one dosing interval at steady state) | up to day 11
Cmax (maximum concentration of metabolite 402 in plasma) | up to day 11
Ae (amount of BILR 355 excreted in the urine over the time interval from 0 to the time of the last urine collection interval) | up to day 11
Metabolite BILR 402 Ae (amount of BILR 402 excreted in the urine over the time interval from 0 to the time of the last urine collection interval) | up to day 11
Number of subjects with adverse events | up to 42 days